CLINICAL TRIAL: NCT03896373
Title: Role of the Neonatal Fc Receptor for IgG in the Pathophysiology of Lupus
Acronym: RFPL
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI18/RFPL; 2019-A00394-53 (Other: IdRCB)
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lupus erythematosus: Patients with inactive lupus erythematosus, active lupus erythematosus or newly diagnosed
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples

SUMMARY:
This study evaluates the expression of the neonatal fc receptor (FcRn) in white blood cells and antigen-presenting cells (APC) in active lupus patients compared to inactive lupus patients and control to investigate if it's upregulated or not.

DETAILED DESCRIPTION:
FcRn is an intracellular receptor which binds the Fc of immunoglobulins G (IgG) and albumin which induce an upgraded half-life of this two proteins.

It's extended role involve the regulation of immune complexes and anti-tumoral immunity, some studies showing a direct correlation between it's expression and the tumor surface and prognosis.

Recently a role in the upregulation of humoral response with a increase of the antibodies's diversity and a more efficient priming of lymphocyte B have been evocated.

The lupus erythematosus is an auto-immune disease mediated by IgG and immune complexes characterized by a high diversity of autoantibodies and a large dysregulation of the immune system in all it's components.

In this study, by analogy with the founding in anti-tumoral immunity, the investigators hypothesised that in an active lupus disease the expression of FcRn is upregulated in the white blood cells and in APC.

This is followed by an extended half life of IgG autoantibodies and immune complexes inducing direct damages by their deposit in tissues and indirectly by upregulating the humoral response, leading to anormal production of a large panel of autoantibodies.

ELIGIBILITY:
Inclusion criteria:

* Lupus erythematosus newly diagnosed or active
* Inactive lupus erythematosus
* Needing a blood sample for diagnosis or follow up
* Signed informed consent

Exclusion criteria:

* Other auto immune disease
* Pregnant or brest feeding
* Legal protection or protected adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient included are hospitalised in the university hospital of Tours in France
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-10-18 (Actual); Study Completion 2020-10-18 (Actual)

PRIMARY OUTCOMES:
Expression of FcRn in active or newly diagnosed lupus erythematosus compared with inactive lupus erythematosus | At baseline
  Measurement in flow cytometry of the fluorescence's mean of FcRn in each type of white blood cells

SECONDARY OUTCOMES:
FcRn genotyping (FCGRT) | At baseline
  FcRn gene polymorphism analysis (FCGRT)
IGHG1 genotyping | At baseline
  IGHG1 gene polymorphism analysis
Expression of FcRn in CD16 monocytes | At baseline
  CD16 is used to differentiate subpopulation of monocytes. The investigators will evaluate the correlation between expression of CD16 and the fluorescence's mean of FcRn measured in flowcytometry.
  This measure will be done for each population of participants
Expression of FcRn in macrophages | At baseline
  After a positive selection of monocytes obtained from participants, the investigators will measure the fluorescence's mean of FcRn in this cells for each population of participants

CONTACTS AND LOCATIONS:
Overall Officials: Valérie GOUILLEUX, PhD, Study Director — University Hospital, Tours
Locations (2):
- France (2):
  - Internal Medicine Service, University Hospital, Tours, Tours
  - Nephrology Service, University Hospital, Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided